CLINICAL TRIAL: NCT03075696
Title: A Multicenter, Open-label, Phase I/II Study to Evaluate the Safety, Efficacy, Tolerability and Pharmacokinetics of Escalating Doses of Glofitamab (RO7082859) as a Single Agent and in Combination With Obinutuzumab Administered After a Fixed, Single Dose Pre-treatment of Obinutuzumab (Gazyva®/Gazyvaro™) in Patients With Relapsed/Refractory B-cell Non-hodgkin's Lymphoma
Brief Title: A Dose Escalation Study of Glofitamab (RO7082859) as a Single Agent and in Combination With Obinutuzumab, Administered After a Fixed, Single Pre-treatment Dose of Obinutuzumab in Participants With Relapsed/Refractory B-cell Non-hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP30179; 2016-001185-28 (EudraCT Number); 2023-505625-14-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2017-03-07; First posted 2017-03-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — glofitamab; obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I: Dose Escalation (Experimental): Participants (single participant cohorts) will receive obinutuzumab pretreatment (Gpt) 1000 milligrams (mg) single dose IV infusion on Day -7 followed by glofitamab IV infusion on Day 1 and Day 8 of Cycle 1. From Cycle 2 onwards, ascending doses of glofitamab will be administered on Day 1 of every 2 week (Q2W) cycle up to Cycle 12 (24 weeks) or until unacceptable toxicity or disease progression. Glofitamab dosing will be initiated at 5 micrograms (mcg) (flat dose) followed by doses of 15 mcg, 45 mcg, 135 mcg, 405 mcg and 810 mcg.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab
- Part II: Dose Escalation (Experimental): In each treatment regimen, participants will receive Gpt 1000 mg IV infusion on Day -7; or 2000 mg either administered on Day -7, or split into two 1000 mg doses on Days -1 and -7. The first glofitamab IV infusion will be given on Day 1 of Cycle 1 and a total of 12 cycles will be administered.
  Monotherapy, glofitamab as a single agent: ascending doses of glofitamab administered on Day 1 of Q2W or every 3 week (Q3W) cycle until either the MTD/OBD is defined.
  Combination Therapy: From Cycle 2 onwards, a fixed dose of 1000 mg obinutuzumab will be administered via IV infusion in combination with ascending doses of glofitamab on Day 1 of Q3W cycle until either the MTD/OBD is defined.
  Step-up dosing: Q3W, participants will receive an initial low dose of glofitamab on Cycle 1 Day 1, followed by a higher dose on Cycle 1 Day 8; the total dose in Cycle 1 will not exceed the previously determined MTD. Higher doses may be explored from Cycle 2 or later cycles.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab
- Part III: Dose Expansion (Experimental): Part III will start once MTD/OBD is defined. Participants will receive Gpt 1000 mg single dose IV infusion on Day -7, followed by glofitamab at a fixed dose regimen or step-up dose regimen on a Q2W or Q3W dosing schedule as determined in Part II. A total of 12 cycles will be administered.
  Combination Therapy: From Cycle 2 onwards, a fixed dose of 1000 mg obinutuzumab will be administered via IV infusion in combination with glofitamab at the dosing regimen determined in Part II.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered at a dose and as per the schedule specified in the respective arms.
  Other Names: RO7082859
Drug: Obinutuzumab — Obinutuzumab 1000 mg single dose IV infusion on Day -7; or 2000 mg single dose administered on Day -7, or split into two 1000 mg doses administered on Days -1 and -7, and per the schedule specified in the respective arms.
  Other Names: RO5072759, GA101, Gazyva®, Gazyvaro™
Drug: Tocilizumab — Tocilizumab will be administered as an IV infusion, if required, for the management of severe Cytokine Release Syndrome (CRS) occurring during or after any infusion of glofitamab, as per the methods described in the Summary of Product Characteristics (SmPC) or other similar local prescribing documents.
  Other Names: Actemra®, Roactemra®

SUMMARY:
This is a Phase I/II, multicenter, open-label, dose-escalation study designed to evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of a novel T-Cell bispecific (TCB), glofitamab, administered by intravenous (IV) infusion as a single agent and in combination with obinutuzumab, following pre-treatment with a one-time, fixed dose of obinutuzumab. This entry-into-human (EIH) study is divided in 3 parts: dose escalation (Parts I and II) and dose expansion (Part III). Single-participant dose-escalation cohorts will be used in Part I, followed by conversion to multiple participant dose-escalation cohorts (Part II), in order to define a tentative maximum tolerated dose (MTD) or optimal biological dose (OBD). The expansion cohorts (Part III) will be initiated when the tentative MTD/OBD is defined, to further evaluate the safety, PK and therapeutic activity of glofitamab.

ELIGIBILITY:
Inclusion Criteria:

* Depending upon study part, a history or status of: 1) a histologically-confirmed hematological malignancy that is expected to express cluster of differentiation (CD)20; 2) relapse after or failure to respond to at least one prior treatment regimen; and 3) no available treatment options that are expected to prolong survival (e.g., standard chemotherapy or autologous stem cell transplant [ASCT])
* Measurable disease, defined as at least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension
* Able to provide a tumor tissue pretreatment biopsy at last relapse or during screening from a safely accessible site, per investigator determination, providing the patient has more than one measurable target lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of >/=12 weeks
* AEs from prior anti-cancer therapy must have resolved to Grade less than or equal to (</=) 1
* Adequate liver, hematological and renal function
* Negative serologic or polymerase chain reaction (PCR) test results for acute or chronic Hepatitis B virus (HBV) infection
* Negative test results for Hepatitis C virus (HCV) and human immunodeficiency virus (HIV)
* Negative serum pregnancy test within 7 days prior to study treatment in women of childbearing potential. Women who are not of childbearing potential who are considered to be post-menopausal (at least 12 months of non-therapy amenorrhea) or surgically sterile (absence of ovaries and/or uterus) are not required to have a pregnancy test

Exclusion Criteria:

* Inability to comply with protocol mandated hospitalizations and restrictions
* Participants with chronic lymphocytic leukemia (CLL), Burkitt lymphoma and lymphoplasmacytic lymphoma
* Participants with a known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Participants with acute bacterial, viral, or fungal infection at baseline, confirmed by a positive blood culture within 72 hours prior to obinutuzumab infusion or by clinical judgment in the absence of a positive blood culture
* Participants with known active infection, or reactivation of a latent infection, whether bacterial, viral, fungal, mycobacterial, or other pathogens or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of dosing
* Prior treatment with systemic immunotherapeutic agents, including, but not limited to, radio-immunoconjugates, antibody-drug conjugates, immune/cytokines and monoclonal antibodies (e.g., anti-cytotoxic T-lymphocyte-associated protein 4 [anti-CTLA4], anti-programmed death 1 [anti-PD1] and anti-programmed death ligand 1 [anti-PDL1]) within 4 weeks or five half-lives of the drug, whichever is shorter, before obinutuzumab infusion on Cycle 1 Day -7
* History of treatment-emergent immune-related AEs associated with prior immunotherapeutic agents
* Documented refractoriness to an obinutuzumab-containing regimen
* Treatment with standard radiotherapy, any chemotherapeutic agent, or treatment with any other investigational anti-cancer agent, including chimeric antigen receptor therapy (CAR-T) within 4 weeks prior to obinutuzumab infusion
* Prior solid organ transplantation
* Prior allogeneic stem cell transplantation (SCT)
* Autologous SCT within 100 days prior to obinutuzumab infusion
* Participant with history of confirmed progressive multifocal leukoencephalopathy (PML)
* Current or past history of central nervous system (CNS) lymphoma
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Participants with a past history of stroke that have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits are allowed
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders and known autoimmune diseases
* Participants with another invasive malignancy in the last 2 years (with the exception of basal cell carcinoma and tumors deemed by the Investigator to be of low likelihood for recurrence)
* Significant or extensive history of cardiovascular disease such as New York Heart Association Class III or IV or Objective Class C or D cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina
* Administration of a live, attenuated vaccine within 4 weeks before obinutuzumab infusion or anticipation that such a live attenuated vaccine will be required during the study
* Received systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within two weeks prior to obinutuzumab infusion. Treatment with corticosteroid </= 25 mg/day prednisone or equivalent is allowed. Inhaled and topical steroids are permitted
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus, erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Participants with a remote history of, or well controlled autoimmune disease, may be eligible to enroll after consultation with the Medical Monitor
* In Part III diffuse large B-cell lymphoma (DLBCL) dexamethasone cohort, participants with a history of hypersensitivity to dexamethasone or systemic corticosteroids will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Part I and II: Percentage of Participants With Dose Limiting Toxicities (DLTs) | From Baseline up to 4 weeks
Part I, II and III: Percentage of Participants With Adverse Events (AEs) | From Baseline up to 90 days after last dose of study drug or until study completion or participant withdrawal (up to 5 years)
Part II: MTD or OBD of Glofitamab | From Baseline up to 4 weeks
Part II: Recommended Phase II Dose (RP2D) of Glofitamab | From Baseline up to 5 years
Part III: Complete Response (CR) Rate as Assessed by Independent Review Committee (IRC) According to Standard Non-hodgkin's Lymphoma (NHL) Response Criteria (Lugano Classification) | From treatment start up to 5 years
Part I, II and III: Area Under the Serum Concentration Versus Time Curve (AUC) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 to Day 71
Part I, II and III: Maximum Serum Concentration (Cmax) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 to Day 198
Part I, II and III: Minimum Serum Concentration (Cmin) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 up to Day 198
Part I, II and III: Clearance (CL) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 to Day 71
Part I, II and III: Volume of Distribution at Steady-state (Vss) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 to Day 71
Part I, II and III: Half-life (t1/2) of Glofitamab | At pre-defined intervals from Cycle 1 Day 1 to Day 71

SECONDARY OUTCOMES:
Part I, II and III: Cmax of Obinutuzumab | Pre-dose of obinutuzumab on Day -7; pre-dose (Hr 0) of glofitamab on Day 1 of Cycle 1
Part I, II and III: Cmin of Obinutuzumab | Pre-dose of obinutuzumab on Day -7; pre-dose (Hr 0) of glofitamab on Day 1 of Cycle 1
Part I, II and III: Anti-drug Antibodies (ADA) to Glofitamab | Pre-dose of obinutuzumab on Day -7; pre-dose (Hr 0) of glofitamab on Day 1 of each cycle from Cycle 2 onwards for a maximum of 8-12 cycles, and at EOT/follow-up visit (up to 5 years)
Parts I and II: Percentage of Participants With Overall Response (Partial Response [PR] or Complete Response [CR]) as Determined by the Lugano Classification | From Baseline up to end of study or discontinuation due to disease progression (up to 5 years)
Part I, II and III: Percentage of Participants With PR or CR (Overall Response Rate [ORR]) as Determined by the Lugano Classifications | From Baseline up to end of study or discontinuation due to disease progression (up to 5 years)
Part I, II and III: Duration of Response (DOR) as Determined by the Lugano Classification | From first occurrence of documented objective response until disease progression, relapse or death due to any cause (up to 5 years)
Part I, II and III: Duration of Complete Response (DOCR) as Determined by the Lugano Classification | From the first occurrence of a documented, complete response, until the time of relapse or death from any cause (up to 5 years)
Part I, II and III: Progression-Free Survival (PFS) as Determined by the Lugano Classification | From first study treatment to the first occurrence of disease progression or death due to any cause (up to 5 years)
Overall Survival (OS) | From the time of first study treatment to death from any cause (up to 5 years)
Time to First Overall Response (TFOR) | From time of treatment start to first documented response (up to 5 years)
Time to First Complete Response (TFCR) | From treatment start to first documented complete response (up to 5 years)
Part III: Health Related Quality of Life (HRQoL) as Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core 30 (EORTC QLQ-C30) | From baseline through follow-up or until disease progression (up to 5 years)
Part III: HRQoL as Assessed by the Functional Assessment of Cancer Therapy-lymphoma (FACT-lym) Scale | From baseline through follow-up or until disease progression (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (8):
  - Ingalls Memorial Hospital, Harvey, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - MSKCC, New York, New York
  - Allegheny Health Network (Pittsburg PA), Pittsburgh, Pennsylvania
  - Hunstman Cancer Institute, Salt Lake City, Utah
  - Swedish Cancer Inst., Seattle, Washington
- Australia (2):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Vseobecna Fakultni Nemocnice v Praze, I. Interni Klinika - Klinika Hematoonkologie VFN a 1. LF UK, Prague, Czechia
- Rigshospitalet, København Ø, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- France (5):
  - Hopital Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - CHU Saint Eloi, Montpellier
  - Ch Lyon Sud, Pierre-Bénite
  - CHU DE RENNES - CHU Pontchaillou, Rennes
- Italy (4):
  - AUSL della Romagna, Ravenna, Emilia-Romagna
  - Fond. IRCCS Istituto Nazionale Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette, Turin, Piedmont
- Auckland Cancer Trial Centre, Auckland, New Zealand
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Centrum Onkologii-Instytut im. M. Sklodowskiej-Curie, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Duran i Reynals L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Univ. 12 de Octubre, Madrid
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan Universtiy Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Phillips TJ, Carlo-Stella C, Morschhauser F, Bachy E, Crump M, Trneny M, Bartlett NL, Zaucha J, Wrobel T, Offner F, Humphrey K, Relf J, Filezac de L'Etang A, Carlile DJ, Byrne B, Qayum N, Lundberg L, Dickinson M. Glofitamab in Relapsed/Refractory Mantle Cell Lymphoma: Results From a Phase I/II Study. J Clin Oncol. 2025 Jan 20;43(3):318-328. doi: 10.1200/JCO.23.02470. Epub 2024 Oct 4. PMID 39365960
- [Derived] Dickinson MJ, Carlo-Stella C, Morschhauser F, Bachy E, Corradini P, Iacoboni G, Khan C, Wrobel T, Offner F, Trneny M, Wu SJ, Cartron G, Hertzberg M, Sureda A, Perez-Callejo D, Lundberg L, Relf J, Dixon M, Clark E, Humphrey K, Hutchings M. Glofitamab for Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2022 Dec 15;387(24):2220-2231. doi: 10.1056/NEJMoa2206913. Epub 2022 Dec 11. PMID 36507690
- [Derived] Frances N, Bacac M, Bray-French K, Christen F, Hinton H, Husar E, Quackenbush E, Schafer M, Schick E, Vyver AV, Richter WF. Novel in Vivo and in Vitro Pharmacokinetic/Pharmacodynamic-Based Human Starting Dose Selection for Glofitamab. J Pharm Sci. 2022 Apr;111(4):1208-1218. doi: 10.1016/j.xphs.2021.12.019. Epub 2021 Dec 22. PMID 34953862
- [Derived] Broske AE, Korfi K, Belousov A, Wilson S, Ooi CH, Bolen CR, Canamero M, Alcaide EG, James I, Piccione EC, Carlile DJ, Dimier N, Umana P, Bacac M, Weisser M, Dickinson M. Pharmacodynamics and molecular correlates of response to glofitamab in relapsed/refractory non-Hodgkin lymphoma. Blood Adv. 2022 Feb 8;6(3):1025-1037. doi: 10.1182/bloodadvances.2021005954. PMID 34941996
- [Derived] Hutchings M, Morschhauser F, Iacoboni G, Carlo-Stella C, Offner FC, Sureda A, Salles G, Martinez-Lopez J, Crump M, Thomas DN, Morcos PN, Ferlini C, Broske AE, Belousov A, Bacac M, Dimier N, Carlile DJ, Lundberg L, Perez-Callejo D, Umana P, Moore T, Weisser M, Dickinson MJ. Glofitamab, a Novel, Bivalent CD20-Targeting T-Cell-Engaging Bispecific Antibody, Induces Durable Complete Remissions in Relapsed or Refractory B-Cell Lymphoma: A Phase I Trial. J Clin Oncol. 2021 Jun 20;39(18):1959-1970. doi: 10.1200/JCO.20.03175. Epub 2021 Mar 19. PMID 33739857